CLINICAL TRIAL: NCT02524353
Title: Follow-up Study of Functional Capacity and Respiratory Muscle Strength in Patients Undergoing Cardiac Surgery
Brief Title: Follow-up Study of Patients Undergoing Cardiac Surgery
Acronym: Follow-up01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Universitário de Votuporanga (Other)
Responsible Party: Principal Investigator, Fernanda Menezes de Siqueira Santana Alves, Fernanda Menezes de Siqueira santana alves, Centro Universitário de Votuporanga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNIFEV01
Record Dates: First submitted 2015-08-11; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery
Keywords: cardiac surgery
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cardiac surgery (Experimental): cardiac surgery
  Interventions: Other: cardiac surgery

INTERVENTIONS:
Other: cardiac surgery — Surgical cardiac procedures despite benefiting the clinical condition of the patient with potential increased survival and reduced risk of death can cause both immediate and long-term functional changes that may influence the appropriate re-inclusion of this individual the daily life practices as well as labor and social activities. Such changes resulting from surgical procedures in the short term are already well documented but the occurrence of these same changes in the late period and its influence on patient's daily lives are not well documented.

SUMMARY:
Countless studies are performed to quantify the severity of heart disease and its influence on the respiratory system, checking that their heart conditions and the surgical process determine pulmonary complications, one of the most common causes of morbidity and mortality in the postoperative period of cardiac surgery . After surgical procedures, there is a reduction of the residual volume (RV), total lung capacity (TLC), vital capacity (VC) and functional residual capacity (FRC), leading to the formation of atelectasis, with alterations in the ventilation-perfusion ( V / Q), the partial pressure of carbon dioxide in arterial blood (PaCO2) and partial pressure of oxygen in arterial blood (PaO 2).

Pulmonary function is impaired in the postoperative period of cardiac surgery, due to various factors common to this major surgery that will drive the patient to develop respiratory complications such as atelectasis and pneumonia. Physical therapy plays an important role in the treatment of patients undergoing cardiac surgery, both in the preoperative period and postoperative, in order to prevent or minimize the respiratory complications.

Follow-up studies on cardiac rehabilitation quantify the quality of all the activities necessary to ensure to patients with heart disease patients the best physical , mental and social conditions so that consequently they are able , with its effort to regain a normal position in the community and lead a active and productive life over time, therefore, the clinical changes resulting from an extensive cardiac surgery are already highly dedicated described in literature but which daily life factors or rehabilitation interventions that the patient will take in the late postoperative period that really assisted in his complete recovery and inclusion into society they are still not well elucidated , so it is appropriate to carry out this project due to the fact exposed to up.

The project to be developed whose main justification clarify issues related to the return or preservation of the individual feature that undergoes extensive cardiac procedure , as well as incidence of mortality after 12 months of the procedure. The current literature does not expressed clearly, possible impacts on functionality and return the daily activities of the individual in the late postoperative period , since such malfunctions in the immediate post operative period are already fully understood.

DETAILED DESCRIPTION:
Will be held during the period from August to November 2015, quantitative descriptive transversal study with patients in the late postoperative period and who underwent cardiac surgery in a hospital of medium complexity in state of sao paulo , Brazil in the period to one year of the procedure. Patients will be recruited via contact by phone to attend in place with certain pre scheduled time for carrying out assessments relevant to the study.

Evaluations shall be performed in hospital in predetermined track, under the sun and accompanied by the examiners. All individuals will be properly oriented and participate in the activities after signing the informed consent (Informed Consent and Informed).

Will be held primarily refers to report cards and progress retroactive filled by students physiotherapy course that evaluated the functional condition and respiratory muscle strength of these individuals included in the study at the time of hospital discharge in cardiac surgical post (last year). The purpose of the consultation of these records is to determine the functional clinical characteristics of these individuals soon after surgery to corroborate the results of these same tests in these patients one year after participants' surgery as well being able to quantify the influence of a number of situations that occurred in the lives of these individuals who may modify in any way the current situation both clinical and social thereof. These evaluation sheets are filed at the physiotherapy clinic.

After consulting retroactive chips, a full interview will be held with the participant, assessing quality of life through specific scores (SF-36), evaluation of daily living habits, social life, work life, independence, recurrent admissions this the participation period of rehabilitation programs and cease habits like smoking, drinking and physical inactivity.

The clinical trials will be conducted: quantification of inspiratory and expiratory muscle strength through the determination of maximal inspiratory pressure (MIP.) And maximal expiratory pressure (MEP.) Using the device which measures and submaximal functional testing through the application of Walk Test 6 minutes (TC6').

The patient will be taken to the track to be traveled for the test and hemodynamic data were to be collected at rest, during and after the test are: blood pressure, heart rate, oxygen saturation.

The patient should be instructed to walk as fast as you can without running, as recommended by the American ThoracicSociety, on a track of 30 meters, marked every 3 meters, with the turning point. By completing the six minutes, the patient should stop immediately. In this way it will be measured the total distance covered by the patient and again all variables at the time of arrest.

The parameters checked during the whole test should be noted , as the distance traveled in meters.

At the end of quantification of clinical and epidemiological data, previous history and current data comparison will be made in order to determine the physical and functional characteristics of these patients in monitoring the late postoperative period .

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamic stability during the tests to be performed
* Post surgical period of one year,
* The level of awareness and appropriate collaboration for instructions and commanding voice and no weakness in the march.
* The surgeon responsible for the surgical procedure the patient must sign a statement authorizing the patient to participate in the study by answering the interview and conduct the walk test.

Exclusion Criteria:

* Need for interruption of fatigue by tests
* Dyspnea,
* Exercise intolerance proposed
* Pains of any kind or expressed will of the patient to stop the activities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of functional capacity in cardiac surgery through the six-minute walk test | 3 months
  Evaluate the postoperative function of patients undergoing cardiac surgery.

SECONDARY OUTCOMES:
quality of life through the SF - 36 (The Short Form (36) Health Survey) | 3 months
  Determine the impact of intrinsic and extrinsic factors related to the surgical procedure that impact the quality of life of long-term individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa, Votuporanga, São Paulo, Brazil

REFERENCES:
- [Background] AlOtaibi KD, El-Sobkey SB. Spirometric values and chest pain intensity three days post-operative coronary artery bypass graft surgery. J Saudi Heart Assoc. 2015 Jul;27(3):137-43. doi: 10.1016/j.jsha.2015.02.002. Epub 2015 Feb 14. PMID 26136627
- [Background] Lizak MK, Nash E, Zakliczynski M, Sliwka J, Knapik P, Zembala M. Additional spirometry criteria predict postoperative complications after coronary artery bypass grafting (CABG) independently of concomitant chronic obstructive pulmonary disease: when is off-pump CABG more beneficial? Pol Arch Med Wewn. 2009 Sep;119(9):550-7. PMID 19776699
- [Background] Johnson D, Kelm C, Thomson D, Burbridge B, Mayers I. The effect of physical therapy on respiratory complications following cardiac valve surgery. Chest. 1996 Mar;109(3):638-44. doi: 10.1378/chest.109.3.638. PMID 8617070
- [Background] Szyca R, Leksowski K. Assessment of patients' quality of life after haemorrhoidectomy using the LigaSure device. Wideochir Inne Tech Maloinwazyjne. 2015 Apr;10(1):68-72. doi: 10.5114/wiitm.2015.49672. Epub 2015 Mar 10. PMID 25960796
- [Background] Sobrinho MT, Guirado GN, Silva MA. Preoperative therapy restores ventilatory parameters and reduces length of stay in patients undergoing myocardial revascularization. Rev Bras Cir Cardiovasc. 2014 Apr-Jun;29(2):221-8. doi: 10.5935/1678-9741.20140021. PMID 25140472
- [Background] Barbalho-Moulim MC, Miguel GP, Forti EM, Campos Fdo A, Costa D. Effects of preoperative inspiratory muscle training in obese women undergoing open bariatric surgery: respiratory muscle strength, lung volumes, and diaphragmatic excursion. Clinics (Sao Paulo). 2011;66(10):1721-7. doi: 10.1590/s1807-59322011001000009. PMID 22012043
- [Background] Tenorio LH, Santos AC, Camara Neto JB, Amaral FJ, Passos VM, Lima AM, Brasileiro-Santos Mdo S. The influence of inspiratory muscle training on diaphragmatic mobility, pulmonary function and maximum respiratory pressures in morbidly obese individuals: a pilot study. Disabil Rehabil. 2013;35(22):1915-20. doi: 10.3109/09638288.2013.769635. Epub 2013 May 7. PMID 23651130
- [Background] Casali CC, Pereira AP, Martinez JA, de Souza HC, Gastaldi AC. Effects of inspiratory muscle training on muscular and pulmonary function after bariatric surgery in obese patients. Obes Surg. 2011 Sep;21(9):1389-94. doi: 10.1007/s11695-010-0349-y. PMID 21229331
- [Background] Graetz JP, Zamuner AR, Moreno MA. Evaluation of maximal inspiratory and sniff nasal inspiratory pressures in pre- and postoperative myocardial revascularization. Rev Bras Cir Cardiovasc. 2012 Dec;27(4):607-13. doi: 10.5935/1678-9741.20120103. PMID 23515734
- [Result] Leggett LE, Hauer T, Martin BJ, Manns B, Aggarwal S, Arena R, Austford LD, Meldrum D, Ghali W, Knudtson ML, Norris CM, Stone JA, Clement F. Optimizing Value From Cardiac Rehabilitation: A Cost-Utility Analysis Comparing Age, Sex, and Clinical Subgroups. Mayo Clin Proc. 2015 Aug;90(8):1011-20. doi: 10.1016/j.mayocp.2015.05.015. Epub 2015 Jul 3. PMID 26149321